CLINICAL TRIAL: NCT06806631
Title: The Effect of Nurse-led Video-assisted Discharge Training on Anxiety and Readiness for Discharge
Brief Title: The Effect of Nurse-led Video-assisted Discharge Training on Anxiety and Readiness for Discharge After Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, HATİCE DEMİRDAĞ, Phd, Uskudar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: do362957
Record Dates: First submitted 2025-01-22; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Discharge Readiness; Nursing; Training
Keywords: anxiety; discharge readiness; discharge training; nursing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Quasi experimental controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video assisted discharge training group (Experimental): The researchers developed a training content by utilizing various sources and consulting expert opinions. DISCERN (quality criteria for consumer health information) tool was used to evaluate the information quality of the educational content and 5 expert opinions were obtained and the educational content was finalized in line with the suggestions. The training content included the problems that patients may experience in the postoperative period, postoperative interventions (movement, breathing and cough exercises), control times, nutrition, do's and don'ts and other nursing care issues. The content of the training video prepared according to the DISCERN scale was found to be sufficient. The training content was then converted into a video training given by the nurse researcher.
  Interventions: Other: Video assisted discharge training
- Control group (No Intervention): Patients will receive routine discharge training in the clinic.

INTERVENTIONS:
Other: Video assisted discharge training — The researchers developed a training content by utilizing various sources and consulting expert opinions. DISCERN (quality criteria for consumer health information) tool was used to evaluate the information quality of the educational content and 5 expert opinions were obtained and the educational content was finalized in line with the suggestions. The training content included the problems that patients may experience in the postoperative period, postoperative interventions (movement, breathing and cough exercises), control times, nutrition, do's and don'ts and other nursing care issues. The content of the training video prepared according to the DISCERN scale was found to be sufficient. The training content was then converted into a video training given by the nurse researcher.
  Arms: Video assisted discharge training group

SUMMARY:
This clinical trial aims to evaluate the effect of nurse-led video-assisted discharge education on discharge readiness and anxiety in patients undergoing coronary artery bypass graft surgery.

The main questions that are aimed to be answered are:

Is there a difference between the discharge readiness levels of patients who received video-assisted discharge training and patients who received classical discharge training?

Is there a difference between the anxiety levels of patients receiving video-assisted discharge training and patients receiving classical discharge training?

Participants:

Experimental group Patients in the intervention group were administered the Readiness for Discharge scale and the State Anxiety Scale on the morning of discharge. Afterwards, the discharge training video prepared by the researchers was sent to their cell phones and they were allowed to watch it with the nurse. The researcher also encouraged the patients to ask questions when they did not understand a topic. Since the video remained on the patient's phone, they could watch it again after discharge. After the training, Discharge Readiness Scale and State Anxiety Scale were administered again.

Control group On the morning of discharge, patients in the control group were administered the Readiness for Discharge Scale and State Anxiety Inventory. The clinic nurse then gave discharge training, which is a clinical routine. After the training, the Readiness for Discharge Scale and State Anxiety Inventory were administered again.

DETAILED DESCRIPTION:
Type of Research This study is a quasi-experimental controlled design. Patients who underwent CABG surgery were divided into 2 groups as patients who received standard discharge training and patients who received video-assisted discharge training.

Place and Sample of the Study The study was conducted between January and October 2023 in a Thoracic-Cardiovascular Surgery Hospital in Istanbul. G*Power version 3.1 was used to calculate the sample size. According to the results of Weiss (2010), the sample size was calculated as 88, 44 intervention and 44 control, with an effect size of 0.32, a significance level (α) of 0.05, an expected power of 0.80, and an effect size estimate of 0.30. The study included 89 patients, 44 in the experimental and 45 in the control groups, who met the inclusion criteria. Inclusion criteria; over the age of 18, good mental health, speak Turkish, have no hearing or vision problems, have had first coronary artery bypass graft surgery.

Data Collection Tools Data were collected using Patient Information Form, Discharge Readiness Scale and State Anxiety Scale.

Patient Information Form: It was prepared by the researchers in line with the relevant literature. The form includes questions about age, gender, marital status, educational status, occupation, place of residence, income status, social security status, presence of an additional disease, smoking, with whom they live at home, presence of a caregiver at home, height, weight, date of hospitalisation, date of surgery, date of discharge.

Discharge Readiness Scale:

The 22-item scale developed by Weiss et al. in 2006 was revised by Weiss et al. in 2014 to consist of eight questions and four subscales (32). It has personal status, knowledge, coping and expected support subscales. The eight questions in the scale are evaluated with scores between 0-10, ranging from low to high. Each measurement is divided into four levels as 9-10 (very high), 8-8.9 (high), 7-7.9 (medium) and <7 (low) (Weiss et al., 2014). The first and second questions measure how the patient feels during the day, the third and fourth questions measure their knowledge about discharge, the fifth and sixth questions measure how and to what extent they can continue their daily life at home after discharge, and the seventh and eighth questions measure the support they can receive at home after discharge (30). The Turkish validity and reliability of this scale developed by Weiss et al. was performed by Kaya et al. in 2017 and the Cronbach α reliability coefficient was found to be 0.74, while this value varied between 0.79-0.93 in subscales (32).

State Anxiety Scale: The scale analyses individuals' state anxiety at a certain time and under a certain condition.

It evaluates how they feel themselves. The scale consists of 20 items with a 4-point Likert-type rating. Scores between 20-80 are obtained from the scale. Higher scores indicate higher anxiety. Internal consistency and reliability of the Turkish form ranged between 0.94 and 0.96 with alpha reliability.38 In this study, the Cronbach's alpha value for the State Anxiety Scale was 0.93, while it was 0.89 for this study.

Intervention The researchers developed a training content by utilising various sources and consulting expert opinions. DISCERN (quality criteria for consumer health information) tool was used to evaluate the information quality of the training content and 5 expert opinions were obtained and the training content was finalised in line with the suggestions. In the training content, the problems that patients may experience in the postoperative period, postoperative interventions (movement, breathing and cough exercises), control times, nutrition, do's and don'ts and other nursing care issues were included. The content of the training video prepared according to the DISCERN scale was found to be sufficient. Then, the training content was converted into a video training given by the nurse researcher.

Collection of data Patients who underwent CABG surgery were informed about the study on the day they came to the clinic and their consent was obtained. The Patient Information Form was first applied to the patients who agreed to participate in the study. Randomisation method was not used to prevent the patients from being affected from each other. The first 44 patients were included in the experimental group and the next 45 patients were included in the control group. Data were obtained using face-to-face interview technique. The information that the patient would be discharged was obtained from the clinic secretary or the nurse working that day.

Experimental group Patients included in the intervention group were administered the Readiness for Discharge Scale and State Anxiety Scale on the morning of discharge. Afterwards, the discharge training video prepared by the researchers was sent to their mobile phones and they were allowed to watch it accompanied by a nurse. The researcher also encouraged the patients to ask questions when they did not understand a topic. Since the video remained on the patient's mobile phone, they could watch it at any time after discharge.

ELIGIBILITY:
Inclusion Criteria:

* First coronary artery bypass graft surgeryi, good mental health, could speak Turkish

Exclusion Criteria:

* had hearing or vision problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Anxiety | Postoperative 30 day
  State anxiety scale score
Discharge readiness | Postoperative 30 day
  Discharge readiness scale score

CONTACTS AND LOCATIONS:
Overall Officials: HATİCE DEMİRDAĞ, Principal Investigator — Üsküdar University
Locations (1):
- Hatice Demirdağ, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No